CLINICAL TRIAL: NCT00318604
Title: Plasma Circulating Deoxyribonucelic Acid (DNA) as a Response Marker
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: 94042
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2006-05-12 (Estimated); Status verified 2006-04

CONDITIONS: Head and Neck Cancer; Esophageal Cancer
Keywords: plasma circulating DNA; hean and neck cancers; esophageal cancer; localized head and neck cancers; localized esophageal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study investigates whether the amount of circulating plasma DNA can be used as a response marker for anti-cancer treatment in treating gross tumors.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancers
* Esophageal cancer
* Undergoing anti-cancer treatments

Exclusion Criteria:

* No distant metastasis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: LeJung Wu, MD, DPhil, Principal Investigator — Far Eastern Memorial Hospital